CLINICAL TRIAL: NCT01676376
Title: A Multi-center, International Study of External Saphenous Vein Support Using eSVS® Mesh in CABG Surgery: The eMESH I Study
Brief Title: The eMESH 1 Feasibility Study
Acronym: eMESH 1
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kips Bay Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11016
Record Dates: First submitted 2012-08-21; First posted 2012-08-30 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Atherosclerosis of Autologous Vein Coronary Artery Bypass Graft(s)
Keywords: CABG; SVG; nitinol mesh; external saphenous vein graft support

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- eSVS Mesh treated saphenous vein graft (Active Comparator): Each subject will be randomized to an eSVS Mesh treated SVG to the right or left coronary system.
  Interventions: Device: eSVS Mesh treated saphenous vein graft
- Control saphenous vein graft (Sham Comparator): Each subject will be randomized to an untreated (no eSVS Mesh) SVG to the right or left coronary system.
  Interventions: Other: Control saphenous vein graft
- Single Vessel Treatment (Active Comparator): Each subject with receive one SVG with eSVS Mesh either to the right or left coronary system.
  Interventions: Device: eSVS Mesh treated saphenous vein graft

INTERVENTIONS:
Device: eSVS Mesh treated saphenous vein graft — During coronary artery bypass graft surgery, one SVG will be randomized to be treated with eSVS Mesh and implanted in the right or left coronary system.
  Arms: Single Vessel Treatment; eSVS Mesh treated saphenous vein graft
Other: Control saphenous vein graft — During coronary artery bypass graft surgery, one SVG will be randomized to be the control (no eSVS Mesh) and implanted in the right or left coronary system.
  Arms: Control saphenous vein graft

SUMMARY:
Multi-center, dual cohort (randomized and single vessel) study designed to demonstrate feasibility, initial safety and performance of the Kips Bay Medical, Inc. eSVS® Mesh as an external vein support device for use over saphenous vein grafts during coronary artery bypass surgery. In the Randomized Cohort, each study subject will receive a SVG without Mesh (control) and a SVG with the eSVS Mesh (treatment). In the Single Vessel Cohort, each study subject will receive one SVG with the eSVS Mesh.

ELIGIBILITY:
Inclusion Criteria:

* Randomized Cohort: Requires CABG surgery with a SVG to the right coronary artery (RCA) system AND the left circumflex artery (LCX) system with a ≥ 70% stenosis in each of the two systems.
* Single Vessel Cohort: Requires CABG surgery with a SVG to the RCA system or the LCX system with a > 70% stenosis in the system.
* Medial sternotomy with cardiopulmonary bypass (CPB) during surgery.
* Both saphenous vein graft length are adequate for planned intervention, vein outer diameter is between 3.6 mm and 7.0 mm and double wall thickness less than 1.4 mm.
* Agreement to post-procedure follow-up contact and testing (including follow-up coronary angiogram).

Exclusion Criteria:

* Concomitant non-CABG cardiac procedure.
* Prior cardiac surgery (does not include percutaneous procedures).
* Cerebrovascular or transient ischemia attack within 30 days of the CABG procedure.
* Age > 85 years.
* Left ventricular ejection fraction ≤ 35%.
* Creatinine > 133 μmol/L (1.5 mg/dL) prior to CABG procedure or on chronic dialysis.
* STEMI within 7 days or total CK > 2 times the upper limit of normal prior to the CABG procedure.
* Both enrolled grafts will feed non-viable myocardial territory.
* Diffuse atherosclerotic disease (> 70%) distal to either of the enrolled target coronary arteries.
* Randomized Cohort: By visual estimate, the target coronary artery diameter of both the right coronary system and left circumflex system must be within 1.5mm of each other.
* Planned endarterectomy of the target coronary artery.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
MACE | 30 days
  The rate of major adverse coronary events (MACE) defined as the rate of the composite of total mortality, MI (Q wave and non Q wave), and/or coronary target vessel revascularization (percutaneous coronary intervention or CABG).
SVG patency determined by angiography | 6 months
  Angiographic patency rate of the enrolled grafts defined as < 50% stenosis.
Technical success implanting eSVS Mesh | intra-operative
  Technical success defined as successful placement of the eSVS Mesh on the saphenous vein and surgical implantation of the SVG.

SECONDARY OUTCOMES:
MACCE and mediastinitis | 5 years
  MACE, MACCE, MI and all mortality rates through five years, mediastinitis rate through 6 months.
SVG patency determined by angiography | 6 months
  Angiographic patency rate of the enrolled grafts defined as < 75%.
Plaque burden | 6 months
  Plaque burden of the enrolled grafts as assessed by IVUS imaging (IVUS Sub-Study).

CONTACTS AND LOCATIONS:
Overall Officials: Lars Englberger, MD, Principal Investigator — University of Bern; John Puskas, MD, Principal Investigator — Emory University
Locations (15):
- United States (5):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - Mayo Clinic / St. Mary's Hospital, Rochester, Minnesota
  - The Valley Hospital, Ridgewood, New Jersey
  - Lenox Hill Hospital, New York, New York
- Czechia (3):
  - General University Hospital, Prague
  - Hospital na Homolce, Prague
  - University Hospital Kralovske Vinohrady, Prague
- France (2):
  - C.H.U. Dupuytren, Limoges
  - Bordeaux University Hospital, Pessac
- Italy (2):
  - Lancisi Hospital, Ancona
  - Heart Hospital - G. Monasterio Tuscany Foundation for Health & Research, Massa
- Catharina Ziekenhuis, Eindhoven, Netherlands
- University Hospital of Bern, Bern, Switzerland
- Royal Brompton Hospital, London, United Kingdom